CLINICAL TRIAL: NCT01392456
Title: Patient Satisfaction With the Use of Three Different Systems as Retention for Implant Supported Mandibular Overdentures.
Brief Title: Validation and Cross-Cultural Adaptation of the Romanian Version of Oral Health Impact Profile in Edentulous Adults
Acronym: ROM-OHIP-ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Concordia Dent Srl (Other)
Collaborators: ITI International Team for Implantology, Switzerland (Other)
Responsible Party: Principal Investigator, Corina Marilena Cristache, Dr Corina Marilena Cristache, DMD, PhD, senior lecturer, Concordia Dent Srl
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 507-207; 316/03 & 507-207 (Other Grant/Funding Number: ITI (INTERNATIONAL TEAM FOR IMPLANTOLOGY) 316/03&507-207)
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Severe Atrophy of the Edentulous Mandible
Keywords: OHIP-EDENT, VALIDATION, OVERDENTURE, ROMANIAN

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Retentive Anchor Group (Active Comparator): 23 fully edentulous patients will receive Retentive Anchors (Institute Straumann AG, Basel Switzerland)as retention system for the two implant overdenture.
  Interventions: Procedure: Insertion of two screw type dental implants
- Magnet Group (Active Comparator): 23 fully edentulous patients will receive Magnets (Institute Straumann AG, Basel Switzerland)as retention system for the two implant overdenture.
  Interventions: Procedure: Insertion of two screw type dental implants
- Locator Group (Active Comparator): 23 fully edentulous patients will receive Locator (Institute Straumann AG, Basel Switzerland)as retention system for the two implant overdenture.
  Interventions: Procedure: Insertion of two screw type dental implants

INTERVENTIONS:
Procedure: Insertion of two screw type dental implants — Each patient (of the 69 recruited) will receive 2 screw-type Straumann (Institute Straumann AG, Basel, Switzerland) standard implants Ø4.1 mm, with SLA surface in the canine region of the mandible with an interconnecting line approaching parallelism with the terminal mandibular hinge axis, in a 1-stage non-submerged procedure according to a strict protocol (Weingart D and ten Bruggenkate 2000).
  Other Names: Straumann (Institute Straumann AG, Basel, Switzerland)

SUMMARY:
The aim of the study is:

1. To validate the Romanian translation of OHIP-EDENT (Oral Health Impact Profile in Edentulous Adults), the short form of OHIP (Oral Health Impact Profile) developed by Allen and Locker for edentulous adults. The OHIP questionnaire is an efficient instrument for assessment of OHRQoL - Oral Health-Related Quality of Life.
2. To compare satisfaction of 69 fully mandibular edentulous patients rehabilitated with implant-supported overdentures with three different types of retention: Retentive Anchors, Magnets, Locator.

DETAILED DESCRIPTION:
Fully edentulism can substantially affect oral and general health as well overall quality of life and inappropriate treatment using classical prosthesis may impaired buccal function, increase alveolar bone loss and also is often unsatisfactory for most patients.

Implant-retained dentures provide successful long-term outcomes, particularly when used to rehabilitate the edentulous mandible (Assad et al. 2004; Chan et al. 1995; Davis et al. 1999). Results achievable with such prostheses are well known: the degree of stability, chewing efficiency, and ultimately patient satisfaction exceeds the benefits obtained with conventional denture treatment.

However few studies have addressed the perception of treatments outcomes by patients and is critically important to determine whether there are meaningful differences based on the type of retention used (Retentive Anchors, Magnets, Locator).

OHIP-EDENT (Oral Health Impact Profile in Edentulous Adults), the short form (19 items) of OHIP (Oral Health Impact Profile) detects the impact of oral health in the quality of life of patients who wear total prosthesis and include questions addressing masticatory capacity, pleasure of eating, level of comfort and relationship problems.

This questionnaire is validated in several languages but still not available in Romanian.

Material and methods

1. Linguistic and cultural adaptation:

   Because the OHIP EDENT had not previously been used in Romania, it was piloted to assess the face and content validity within the target population. The OHIP EDENT was linguistically and culturally adapted to our setting by using the back translation technique (according to guidelines provided by Beaton et al. 2000) in order to maintain cross-cultural equivalence. In this procedure, translations were independently made by two bilingual persons, who then discussed and produced a consensus Romanian version (T1 and T2 produced T12), which was translated back into English by two professional English translator (one native English) who had never seen the original version (BT1 and BT2 versions).

   The conceptual equivalence between the original instruments and the back-translated versions was supported by an expert committee (formed by 3 researchers: methodologist, two experts on quality of life studies, and the four translators). The definitive Romanian version was produced after the face and content validity results in the pilot study had been approved by this committee.
2. Pilot study:

   Ethical approval and specific written consent were obtained from the relevant authorities before the pilot study were started.

   The pilot study was conducted in a convenience sample (n=35) obtained from mandibular edentulous patients who came to the Dental School, University of Medicine and Pharmacy Bucharest, Romania and Concordia Dent Clinic, Bucharest. Participants were clinically examined according to the WHO (World Health Organization) methodology and completed the pilot OHIP EDENT.

   The comprehensiveness of the instrument was tested by asking about difficulties in understanding items or frequencies, in order to optimize the face and content validity before the main study.

   Reproducibility was evaluated by measuring test - retest reliability. Test-retest reliability was calculated using intraclass correlation coefficient (ICC). The sample of 35 respondents fully edentulous was interviewed two weeks after the first interview.
3. Main Study:

Patient satisfaction was assessed with the aid of OHIP-EDENT questionnaire validated initial (with the original denture), after 6 months and at 1, 3, 5 years post overdenture insertion.

ELIGIBILITY:
Inclusion Criteria:

* Fully mandibular edentulous patients
* Complains about the stability of the existing mandibular denture satisfactory from a technical point of view.
* Acceptance of a mandibular over-denture retained by two endosseous implants.
* Patients agree to a 5-year follow-up period.

Exclusion Criteria:

* Insufficient bone volume (height and with) for inserting at least a 10 mm implant (Ø 4,1).
* Angle class II relationship.
* Physical severe consideration that will affect the minimal invasive surgical procedure or constitute a hindrance for a 5-year follow-up.
* History of radiotherapy in the head and neck region.
* History of pre-prosthetic surgery (including bone graft procedures) or previous oral implants.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2004-06; Primary Completion 2010-09 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
OHIP-EDENT linguistic and cultural adaptation in Romanian | Two-weeks
  Steps for validation:
  * linguistic and cultural adaptation of the original instrument to Romanian;
  * pilot study to assess face and content validity;
  * main study to assess the reliability and construct validity. OHIP-EDENT questionnaire includes 19-items addressing masticatory capacity, pleasure of eating, level of comfort, and relationship among others while wearing the prosthesis and detects the impact of oral health in the quality of life of edentulous adults wearing total prosthesis. Response categories:4=very often; 3=fairly often; 2=occasionally; 1=hardly ever; 0=never/don't know.

SECONDARY OUTCOMES:
Evaluation of patient satisfaction with the use of three different systems as retention for implant supported mandibular overdentures. | 5 years
  Patient satisfaction is assessed with the use of OHIP-EDENT questionnaire validated in Romanian language.
  The questionnaire is administrated initial (before surgery for assessing patient satisfaction with the original denture), after 6 months of implant over-denture insertion (T) and at 1,3 and 5-year follow-up (T1, T3, T5).
  The means scores will be calculated. Lower scores represents a good perception of the oral conditions, good satisfaction level and good masticatory capacity.

CONTACTS AND LOCATIONS:
Overall Officials: CORINA MARILENA I CRISTACHE, DMD, PhD, Principal Investigator — CONCORDIA DENT CLINIC
Locations (1):
- Concordia Dent Clinic, Bucharest, Romania

REFERENCES:
- [Background] Zani SR, Rivaldo EG, Frasca LC, Caye LF. Oral health impact profile and prosthetic condition in edentulous patients rehabilitated with implant-supported overdentures and fixed prostheses. J Oral Sci. 2009 Dec;51(4):535-43. doi: 10.2334/josnusd.51.535. PMID 20032605
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Assad AS, Abd El-Dayem MA, Badawy MM. Comparison between mainly mucosa-supported and combined mucosa-implant-supported mandibular overdentures. Implant Dent. 2004 Dec;13(4):386-94. doi: 10.1097/01.id.0000144512.43654.08. PMID 15592001
- [Background] Weingart D, ten Bruggenkate CM. Treatment of fully edentulous patients with ITI implants. Clin Oral Implants Res. 2000;11 Suppl 1:69-82. doi: 10.1034/j.1600-0501.2000.011s1069.x. PMID 11168258
- [Background] Chan MF, Johnston C, Howell RA, Cawood JI. Prosthetic management of the atrophic mandible using endosseous implants and overdentures: a six year review. Br Dent J. 1995 Nov 11;179(9):329-37. doi: 10.1038/sj.bdj.4808917. PMID 7495628
- [Background] Davis DM, Packer ME. Mandibular overdentures stabilized by Astra Tech implants with either ball attachments or magnets: 5-year results. Int J Prosthodont. 1999 May-Jun;12(3):222-9. PMID 10635189
- [Background] Naert I, Alsaadi G, Quirynen M. Prosthetic aspects and patient satisfaction with two-implant-retained mandibular overdentures: a 10-year randomized clinical study. Int J Prosthodont. 2004 Jul-Aug;17(4):401-10. PMID 15382775